CLINICAL TRIAL: NCT05876598
Title: BACTERIUM: Study for a Machine-learning-based Model to Predict Bloodstream Infections
Acronym: BACTERIUM
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: BACTERIUM-4407
Record Dates: First submitted 2023-03-16; First posted 2023-05-25 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Infection, Bloodstream
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: antibiotic treatments — The outcome of the study will be to implement Prediction Models to support clinicians for the assessment of risk of having a bloodstream infection.

SUMMARY:
An increase of healthcare-associated infections caused by multidrug- resistant organisms (MRDO) is currently observed. One of the main causes of the emergence of a MDRO infection is an overuse of antibiotics. Therefore, saving useless antibiotic treatment is currently a priority from a public health point of view. The evaluation of the risk of having a bloodstream infection will allow both activating faster treatment decisions (when the risk is significantly high) or to save useless resources in terms of diagnostic tests and treatments, also limiting the potential for side effects (when the risk is significantly low).

ELIGIBILITY:
Inclusion Criteria:

1. adult patients hospitalized at the Gemelli Polyclinic Foundation
2. having at least one performed blood culture
3. starting an antibiotic therapy

Exclusion Criteria:

1. blood cultures with contaminants
2. <18 years old
3. died after less than 48 hours from blood cultures positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients hospitalized at the Gemelli Polyclinic Foundation
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of appropriate antibiotic therapy in patients with bloodstream infections | 24 months
  1) number of patients with bloodstream infections with appropriate antibiotic therapy before and after the application of the predictive model "Bacterium"
Blood cultures | 24 months
  number of blood cultures done before and after the application of the predictive model "Bacterium"

CONTACTS AND LOCATIONS:
Overall Officials: Rita Murri, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Agostino Gemelli Irccs, Rome, Italy

IPD SHARING:
Plan to Share IPD: No